CLINICAL TRIAL: NCT06705218
Title: Changing Mindsets to Improve Whole Patient Health: A Randomized Controlled Trial of a Novel mHealth Intervention for People Diagnosed With Cancer
Brief Title: Exploring Mindsets, Beliefs and Resilience Across the Cancer Experience
Acronym: EMBRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01AT012618 (NIH); R01AT012618 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Mindset; Wellbeing; Resilience; Functioning
MeSH Terms: conditions — Neoplasms | interventions — Stress Mindset Measure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINDSET (Experimental): 2.5-hour mHealth intervention consisting of three modules containing brief films and corresponding interactive reflection activities aimed to improves whole patient health (physical, social, emotional, and functional quality of life as measured by the FACT-G) in patients undergoing systemic treatment for cancer with curative intent. Films feature interviews with people living with cancer describing their experience with diagnosis, treatment, and recovery, and the importance of their mindsets during their experience. The films also feature Stanford faculty with expertise in oncology, psychiatry, and psychology who offer a scientific framework for the importance of mindsets during cancer treatment and provide examples from their clinical practices. The reflection exercises that follow the films are designed to help patients craft a personalized strategy (a) for changing maladaptive mindsets and maintaining adaptive ones and (b) for translating ideas from the film into actionable behavio
  Interventions: Behavioral: MINDSET
- Digital Information Series for Cancer (Active Comparator): This behavioral intervention provides educational information on coping strategies for individuals undergoing cancer treatment through a hybrid of videos and corresponding questions.
  Interventions: Behavioral: Digital Information Series for Cancer

INTERVENTIONS:
Behavioral: MINDSET — 2.5-hour mHealth intervention consisting of three modules containing brief films and corresponding interactive reflection activities aimed to improves whole patient health (physical, social, emotional, and functional quality of life as measured by the FACT-G) in patients undergoing systemic treatment for cancer with curative intent. Films feature interviews with people living with cancer describing their experience with diagnosis, treatment, and recovery, and the importance of their mindsets during their experience. The films also feature Stanford faculty with expertise in oncology, psychiatry, and psychology who offer a scientific framework for the importance of mindsets during cancer treatment and provide examples from their clinical practices. The reflection exercises that follow the films are designed to help patients craft a personalized strategy (a) for changing maladaptive mindsets and maintaining adaptive ones and (b) for translating ideas from the film into actionable behavior
  Arms: MINDSET
Behavioral: Digital Information Series for Cancer — This behavioral intervention provides educational information on coping strategies for individuals undergoing cancer treatment through a hybrid of videos and corresponding questions.
  Arms: Digital Information Series for Cancer

SUMMARY:
The goal of this clinical trial is to test the effect of digitally delivered programs on the health, wellbeing, and functioning of newly diagnosed cancer patients.

Participants will be randomized to one of two digital programs. Both groups are equally important for the study.

Participants will be asked to complete:

* Questionnaires. Answers to the questionnaires will help the investigators understand how participants doing through the study.
* Modules. Participants will receive access to digital courses developed by experts at Stanford University.
* Blood Samples. At home blood collection kits will help the investigators understand how participants' bodies are responding over time. Kits will be sent and returned by mail.

DETAILED DESCRIPTION:
A cancer diagnosis and its subsequent treatment affects whole patient health -- disrupting the full spectrum of physical, social, emotional, and functional quality of life. An estimated 83% of cancer patients report low to very low quality of life. Individuals receiving chemotherapy report experiencing over 13 concurrent symptoms, including fatigue, sleep difficulties, and pain. 30%-40% of people with cancer report significant psychological symptoms, including anxiety and depression. Such disruptions in mental health and quality of life, in turn, exacerbate physical symptoms and can worsen clinical outcomes. Despite growing evidence of the complex, interconnected pathways linking the mind and body, scalable interventions that efficiently target whole-person health upon diagnosis of a life-altering disease such as cancer have not yet been developed. Existing medical treatments, focus on the physiological aspects of the disease. Existing psychological treatments, such as Cognitive Behavior Therapy (CBT) and Mindfulness Based Stress Reduction (MBSR), apply a broad range of cognitive and behavioral strategies to reduce diffuse symptoms of depression and anxiety. Such ancillary programs for psychological care are routinely proposed as methods to reduce distress and symptoms, restore function, and improve quality of life, but they are frequently inaccessible to patients and notoriously difficult to scale. The MINDSET intervention aims to close this major treatment gap and promote whole patient health by targeting patient mindsets at the point of diagnosis. This proposal builds on our extensive foundational research completed over the past 6 years with support of the NIH New Innovator Award (DP2 AT009511) to test a novel mHealth intervention targeting patient mindsets at the point of diagnosis. In our prior research, we showed that a 2.5-hour digital MINDSET intervention significantly improves whole patient health (physical, social, and emotional functioning as measured by the FACT-G) in patients undergoing systemic treatment for cancer with curative intent compared to a Treatment as Usual (TAU) control. Leveraging our interdisciplinary team of experts in oncology, psychology, psychiatry, mHealth, and biostatistics, we aim to expand on this prior research to address this large and costly gap in clinical care. We propose a fully decentralized Phase 3 randomized controlled trial in which 440 cancer patients treated for non-metastatic solid tumors and hematological malignancies will be allocated to either a (1) MINDSET or (2) Matched Attention Control (MAC) condition. Patient-reported primary outcomes (FACT-G Total Score) and secondary outcomes (anxiety, depression, affect, sleep, coping, symptom distress, patient activation/engagement, and inflammatory biology) will be assessed at weeks 0 (baseline), 2, 4, 6, and 10. Durability of the effect of the intervention will be measured at two follow-up timepoints: 3 months, and 6 months after study completion. By promoting health at the psychological, behavioral, and biological levels, MINDSET interventions have the potential to become a highly impactful and complementary tool for promoting whole patient health.

ELIGIBILITY:
Inclusion Criteria:

* Initial (non-recurrent) diagnosis of non-metastatic (stage I-III) or hematological malignancy.
* Diagnosis in the past 150 days.
* Currently receiving active systemic treatment or with a planned systemic treatment (including chemotherapy, immunotherapy or other targeted therapies).
* Eighteen years of age or older.
* Fluent in English.
* Currently reside in the United States.
* Access to a computer, tablet, or smartphone (a mobile phone that performs many of the functions of a computer, typically including a touchscreen interface, internet access, and an operating system capable of running downloaded applications, or tablet that runs iOS or Android software, with cellular data service or wifi access).

Exclusion Criteria:

* Failure to meet inclusion criteria.
* Currently receiving treatment for severe depression, severe anxiety, bipolar disorder, post-traumatic stress disorder, or schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - General (FACT-G) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Physical, emotional, social and functional quality of life will be assessed using the FACT-G questionnaire. The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of quality of life in cancer patients: Physical, social, emotional, and functional well being. Original development and validation involved 854 patients with cancer and 15 oncology specialists.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-A) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Anxiety will be measured using the 8 item Patient-Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-A). The PROMIS-A measures fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart,dizziness). The items in the PROMIS negative affect banks use a 7-day time frame and a 5-point rating scale that ranges from 1 ("Never") to 5 ("Always"), with higher scores indicating greater severity of anxiety symptoms. The standardized T-Score for cancer patients reference population is 50 and the minimally clinically important difference (MCID) in T-scores is 3.0-4.5. Anxiety T-scores can be interpreted categorically as ≤55 = normal; 56-60 = mild; 61-70 = moderate; ≥71 = severe.
Patient-Reported Outcomes Measurement Information System - Depression Short Form 8b (PROMIS-D) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Depression will be measured using the 8 item the Patient-Reported Outcomes Measurement Information System - Depression Short Form 8b (PROMIS-D). The PROMIS-D content focuses on negative mood (sadness, guilt), views of self (self- criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). The items in the PROMIS negative affect banks use a 7-day time frame and a 5-point rating scale that ranges from 1 ("Never") to 5 ("Always"), with higher scores indicating greater severity of depressive symptoms. The standardized T-Score for the cancer patient reference population is 50 and the minimally clinically important difference (MCID) in T-scores is 3.0-4.5. Depression T-Scores can be interpreted categorically as ≤55 = normal; 56-60 = mild; 61-70 = moderate; ≥71 = severe.
Positive and Negative Affect (I-PANAS-SF) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Positive and negative affect will be measured by the International version of the Positive and Negative Affect Schedule-Short Form (PANAS-SF). This is a cross-culturally validated version of the widely affect measure that consists of 10 items; 5 items measuring negative affect and 5 items measuring positive affect.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System - Sleep Disturbance Short Form 8b (PROMIS-Sleep Disturbance) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Sleep disturbance will be measured using the 8 item Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS-Sleep Disturbance). The PROMIS-Sleep Disturbance content focuses on perceptions of sleep quality, sleep depth, and restoration associated with sleep. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
International Physical Activity Questionnaire (IPAQ) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Physical activity will be measured using the 8-tem Short Form of the International Physical Activity Questionnaire (IPAQ). The purpose of the questionnaire is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity by estimating the time spent performing physical activities (moderate to vigorous) and inactivity (time spent sitting).
Coping Behaviors- Cancer Behavior Inventory (CBI) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Coping will be measured using the Cancer Behavior Inventory (CBI). The short version of the CBI is a 12-item measure of self-efficacy for coping with cancer. Items are rated on a 5-point Likert scale indicating confidence in a range of coping skills. The CBI yields a single summary score representing overall confidence in engaging in adaptive coping behaviors.
Patient Activation Measure (PAM-SF) | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  The Patient Activation Measure-Short Form (PAM-SF) is a 13-item measure that assesses patient knowledge, skill, and confidence for self-management.
Rotterdam Symptom Checklist (RSCL)-Physical Symptom Subscale | Treatment Phase: Weeks 0 (Baseline), 2, 4, 6, 10 Follow Up: Months 3, 6
  Symptom distress will be measured using the 25 item physical symptom distress subscale of the Rotterdam Symptom Checklist (RSCL). All items are rated on a 4-point Likert scale ranging from (1) not at all to (4) very much. Higher scores (calculating by taking the sum of the items) are indicative of greater distress or impairment.
Patient Global Impression of Change | Treatment Phase: Weeks 2, 4, 6, 10; Follow Up: Months 3, 6
  The Patient Global Impression of Change is a 3 item measure that assesses a patient's perceived improvement (since the start of the study) across 3 domains: Anxiety, Depression, and Global Wellbeing. Items are rated on a 7-point likert scale from 1 (Very much worse) to 7 (Very much improved).
Inflammatory activity as measured by a MILLIPLEX Human 48 plex (Millipore) | Treatment Phase: Weeks 0 (Baseline), 4, 10 Follow Up: Months 6
  Blood draws will be conducted using at-home blood device such as the Tasso-M20 self-administered home blood sampling method and multiomics testing. The Tasso-M20 device is CE marked and FDA registered. Using the provided kit instructions and contents, subjects will collect the Tasso-M20 blood sample in a self-administered, unsupervised manner which involves attaching the device on their arms for 5 minutes to collect 4 samples of 17.5μLof blood (dry blood spots) (visit Tasso for additional instructions and information) and then ship the device in a pre-labeled envelope back to Stanford where samples will be de-identified and stored in a -80 degree freezer. All de-identified samples will be assayed by the Stanford Human Immune Monitoring Lab (HIMC) using the MILLIPLEX Human 48-plex assay which identifies hormone biomarkers related inflammatory biology.

CONTACTS AND LOCATIONS:
Overall Officials: Alia J Crum, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate clinical trials data from all arms of the study will be available on osf.io, the Open Science Framework (OSF), hosted by the Center for Open Science, along with related metadata. Objectives, hypotheses, methods, and analytic plan will be pre-registered on OSF prior to accessing the study data.
Time Frame: All scientific data generated from this project will be made available at the time of their publication or the end of the funding period, whichever comes first.